CLINICAL TRIAL: NCT07281404
Title: Open-label Lead-in Study of Single-dose 0.7% YASO GEL Followed by a Phase 1 Randomized, Double-blind Dose-escalation Study to Assess Safety and Pharmacokinetics of 2% YASO GEL
Brief Title: FIH Lead-in Study of YASO GEL Followed by a Phase 1 Randomized, Double-blind Study to Assess Safety and Pharmacokinetics of YASO GEL
Acronym: PPCM-01
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yaso Therapeutics Corporation (Industry)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Magee-Women's Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PPCM-01; 1R44HD118927-01 (NIH)
Record Dates: First submitted 2025-12-10; First posted 2025-12-15 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Early-phase Safety and PK Study of a Vaginal Gel
Keywords: Contraceptive activity; HIV prevention; Antimicrobial activity; Sexual activity; Vaginal gel; YASO GEL; Coital exposure; First-in-human; Mucosal drug delivery
MeSH Terms: conditions — Sexual Behavior

STUDY DESIGN:
Intervention Model Description: This first-in-human study consists of three parts. A 6-participant open-label lead-in cohort will receive a single low dose of the investigational contraceptive to assess initial safety and tolerability. The main Phase 1 study is a randomized, double-blind, parallel-group trial enrolling 32 participants, conducted in two stages: Stage 1 participants receive a single full-strength dose with 21-day follow-up, and Stage 2 participants receive daily full-strength doses for 7 days with 28-day follow-up. A 12-participant non-randomized coital sub-study will further assess safety and exploratory endpoints in the context of sexual activity, with and without use of the investigational product. Participants in the randomized Phase 1 portion remain in their assigned intervention arm throughout the study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Lead-in study (Experimental): Participants receive a single low dose of the investigational contraceptive to assess initial safety and tolerability.
  Interventions: Drug: YASO GEL
- Phase 1, Stage 1 - Active Drug (Experimental): Participants receive a single full-strength dose of the investigational contraceptive in a randomized, double-blind design.
  Interventions: Drug: YASO GEL
- Phase 1, Stage 1 - Placebo (Placebo Comparator): Participants receive a single dose of placebo in a randomized, double-blind design.
  Interventions: Drug: Placebo gel
- Phase 1, Stage 2 - Active Drug (Experimental): Participants receive daily full-strength doses of the investigational contraceptive for 7 days in a randomized, double-blind design.
  Interventions: Drug: YASO GEL
- Phase 1, Stage 2 - Placebo (Placebo Comparator): Participants receive daily placebo doses for 7 days in a randomized, double-blind design.
  Interventions: Drug: Placebo gel
- Coital Sub-study (Experimental): Participants receive full-strength investigational contraceptive in an open-label sub-study to further assess safety and exploratory endpoints.
  Interventions: Drug: YASO GEL

INTERVENTIONS:
Drug: YASO GEL — Contraceptive gel
  Arms: Coital Sub-study; Lead-in study; Phase 1, Stage 1 - Active Drug; Phase 1, Stage 2 - Active Drug
Drug: Placebo gel — Inactive placebo gel matching the investigational contraceptive
  Arms: Phase 1, Stage 1 - Placebo; Phase 1, Stage 2 - Placebo

SUMMARY:
The goal of this clinical trial is to assess the safety and pharmacokinetics of YASO GEL in healthy adult participants. This is a first-in-human study designed to understand how the gel is absorbed and distributed in plasma and vaginal fluid, and to evaluate the methods used to measure drug levels in humans.

The main questions the study aims to answer are:

What is the preliminary safety and tolerability of YASO GEL at a subtherapeutic 0.7% dose?

How is YASO GEL absorbed and distributed, and does sexual activity affect its pharmacokinetics?

Participants will:

Receive an application of YASO GEL.

Provide blood and vaginal fluid samples for pharmacokinetic analysis.

Participate in a sub-study evaluating the impact of sexual activity on safety and drug exposure.

Additional information on product acceptability, adherence, and exploratory laboratory analyses will be collected to inform the design of future studies.

DETAILED DESCRIPTION:
This study initiates with a first-in-human lead-in study using a subtherapeutic 0.7% dose of YASO GEL. The study aims to provide a preliminary assessment of PPCM pharmacokinetics in plasma and vaginal fluid, and to validate a bioanalytical assay to be used to measure efficacy in both the Phase 1 and sub studies. Data from this study will help ensure that pharmacokinetic sampling is adequate for subsequent clinical trials and will provide initial safety information to support a Phase 1 study.

The subsequent randomized double-blind Phase 1 study will use a therapeutic 2.0% dose of YASO GEL administered once in Stage 1 of the Phase 1 study and once daily for 7 days in Stage 2 of the Phase 1 study. The Phase 1 study is designed to provide comprehensive baseline safety and pharmacokinetic data in a dose response manner. As such, it is important to assess the genitalia (vulva, perineum and vagina for female participants and penis, scrotum, and perineum for male participants) after each dose for safety, initially with single dose and then with repeated dosing. Because it is anticipated that a coitally-dependent product will be applied prior to each act of coitus, and individuals may have coitus more than once a day, future studies will evaluate more frequent dosing and further characterize the YASO GEL safety profile.

Secondarily, acceptability and adherence data will be collected to inform future product design and patient education. Exploratory endpoints include assessment of vaginal fluid samples for vaginal microbiome, soluble immune mediators, ex-vivo contraceptive activity and anti-microbial activity against both HIV and Ng.

A sub-study is included to evaluate the impact of coitus on safety and pharmacokinetics of YASO GEL use. This study will also collect acceptability and adherence data to inform future product design and patient education. Vaginal fluid samples will be assessed for contraceptive activity and ex vivo anti-microbial activity against both HIV and Ng, in an exploratory fashion to inform future study design.

The study will include healthy adult participants. Female participants will apply the gel internally in all studies. Male participants will apply the gel externally in the Lead-in and Phase 1 studies and be exposed to the gel in the coital sub-study. The results from this study will guide the design of future studies and help establish the safety and efficacy profile of YASO GEL in humans.

ELIGIBILITY:
Inclusion Criteria:

* 4.1.1 Lead-in and Phase 1 Studies

Individuals who meet the following criteria are eligible for inclusion in the study (see additional gender specific criteria at the end of the section):

1. Adults who are:

   * Women aged 18 through 45 years (inclusive)
   * Men aged 18 years and over at Screening
2. Cisgender individuals with no history of gender reassignment impacting hormones or genital anatomy
3. Able to communicate in English
4. Provide written informed consent before any study-related activities are carried out and must be able to understand the full nature and purpose of the trial, including possible risks and adverse effects.
5. Willing and able to comply with all scheduled visits, treatment plans, laboratory tests and other study procedures.
6. Provide adequate locator information (per site SOP)
7. Understand and agree to local STI reporting requirements
8. In general good health, in the opinion of the investigator
9. Agree not to participate in other concurrent interventional and/or drug trials

Female specific criteria:

1. Women ≥ 21 years must have documentation of a satisfactory Pap within the past 3 years consistent with Grade 0 according to the Female Genital Grading Table for Use in Microbicide Studies Addendum 1 (Dated November 2007) to the DAIDS Table for Grading Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017, or satisfactory evaluation with no treatment required of Grade 1 or higher Pap result. If result is not available, Pap test will be performed at screening.
2. Regular menstrual cycles of approximately 21 to 35 days apart with no undiagnosed intermenstrual menstrual bleeding Note: This criterion is not applicable to participants using continuous combination oral contraceptive pills, patches, or progestin-only contraceptive methods (progestin-only pills, depot medroxyprogesterone acetate (DMPA), etonogestrel subdermal implant, or levonorgestrel-releasing IUD), as the absence of regular menstrual cycles and break-through bleeding are common in these contexts.
3. Using an effective method of contraception and intending to continue use of an effective method for the duration of study participation. Acceptable methods are:

   * hormonal methods (except contraceptive vaginal rings)
   * IUD
   * sterilization of participant or partner
   * heterosexual abstinence
   * sexually abstinent for the past 90 days before enrollment and planning to remain abstinent for the duration of study participation
4. Must agree to abstain from insertion of anything other than IP into the vagina or anus (e.g., penis, tongue, finger, sex toy, lubricant, tampon, etc.) for at least 48 hours prior to the Enrollment Visit, the duration of treatment, and at least 48 hours after treatment.

Male specific criteria:

a. Must agree to abstain from:

* Use of any genitally applied products other than IP (except soap/water for general hygiene and study provided condoms for at least 24 hours prior to treatment days and at least 48-hr after treatment
* Masturbation or intercourse (anal, vaginal, or receptive oral) on treatment days and at least 48-hr after treatment

4.1.2 Inclusion Criteria - Sub-Study

Heterosexual couples who meet the following criteria are eligible for inclusion in the study:

Couple-level criteria:

1. Women aged 18 through 45 years (inclusive) and men aged 18 through 55 years (inclusive) at screening
2. Provide written informed consent before any study-related activities are carried out and must be able to understand the full nature and purpose of the trial, including possible risks and adverse effects.
3. Willing and able to comply with all scheduled visits, treatment plans, laboratory tests and other study procedures.
4. Heterosexual couples in a mutually monogamous relationship ≥ 6 months prior to Screening with intent to remain in relationship for duration of study participation
5. Both partners willing to participate and coitally active
6. Cisgender individuals with no history of gender reassignment impacting hormones or genital anatomy
7. Both partners independently report not using barrier contraception and/or barrier protection as part of normal coital routine and report the intent to continue said sexual practice for the duration of study participation
8. Able to communicate in English
9. Provide adequate locator information, as defined in site SOP
10. Must be in general good health in the opinion of the investigator
11. Must agree to not to participate in other concurrent interventional and/or drug trials

Female specific inclusion criteria:

1. Not pregnant or breastfeeding and not planning pregnancy during study participation
2. Women ≥ 21 years must have documentation of a satisfactory Pap within the past 3 years consistent with Grade 0 according to the Female Genital Grading Table for Use in Microbicide Studies Addendum 1 (Dated November 2007) to the DAIDS Table for Grading Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017, or satisfactory evaluation with no treatment required of Grade 1 or higher Pap result. If result is not available, Pap test will be performed at Screening.
3. Regular menstrual cycles of approximately 21 to 35 days apart with no undiagnosed intermenstrual menstrual bleeding Note: This criterion is not applicable to participants using continuous combination oral contraceptive pills, patches, or progestin-only contraceptive methods (progestin-only pills, depot medroxyprogesterone acetate (DMPA), etonogestrel subdermal implant, or levonorgestrel-releasing IUD), as the absence of regular menstrual cycles and break-through bleeding are common in these contexts.
4. Using an effective method of contraception and intending to continue use of an effective method for the duration of study participation. Acceptable methods are:

   * hormonal methods (except contraceptive vaginal rings)
   * IUD
   * Female sterilization
5. Must agree to abstain from use of any vaginal products (e.g., lubricants, feminine hygiene products, sex toys, vaginally administered contraceptive products with the exception of study provided condoms) other than IP for at least 48 hours prior to coital visits and at least 48 hr after coital visits

Male specific inclusion criteria:

1. Must agree to abstain from

   * use of any genitally applied products, except soap/water for general hygiene, for at least 24 hours prior to coital visits and at least 48-hr after coital visits
   * masturbation or intercourse (anal, vaginal, or receptive oral) for 72 hours before each coital visit.
2. Have no history of abnormal sperm or semen abnormality

Exclusion Criteria:

* 4.2.1 Lead-in and Phase 1 Study, as well as the Sub-Study Individuals who meet any of the following criteria will be excluded from the study

General exclusions:

1. Plans to relocate away from the study site area during the period of study participation
2. Genital piercings and/or tattoos
3. Have been diagnosed with genital HSV, with the first occurrence (initial episode) within three months prior to Screening
4. Have had three or more outbreaks of genital HSV within the last year
5. History of recurrent rash/dermatosis (e.g., eczema) in the genital area
6. History of autoimmune disease
7. History of adverse reaction to PPCM, methylparaben, propylparaben, hydroxypropyl methylcellulose (HPMC), or xanthan gum
8. Known HIV seropositivity
9. Non-therapeutic injection drug use in the 6 months prior to Screening
10. Use of HIV PrEP or post-exposure prophylaxis within prior 6 months
11. Use of systemic immunomodulatory medications within the 30 days prior to planned enrollment
12. Participation in another research study involving drugs or medical devices within the 30 days prior to Enrollment
13. Recent use (within last 14 days) and/or unwillingness to abstain from use of vaginally administered medications (including condoms containing Nonoxynol-9 [N-9]) for the duration of the study from enrollment through all follow up visits but not including periods between study phases.
14. Laboratory abnormalities at screening:

    Note: Grade is per Version 2.1 of the DAIDS Toxicity Table
    1. HIV seropositive
    2. Decreased white blood cell count Grade 2 or higher
    3. Hemoglobin Grade 1 or higher
    4. Grade 2 or higher ALT and/or AST (i.e., ≥ 2.5x the site laboratory upper limit of normal [ULN])
    5. Calculated creatinine clearance Grade 2 or higher (i.e., ≤ 90 mL/minute using the Cockcroft-Gault equation.

       * (140 - age in yrs) x (weight in kg) x (0.85)/72 x (serum Cr in mg/dL)

         * (140 - age in yrs) x (weight in kg)/72 x (serum Cr in mg/dL)
15. Symptomatic and/or clinical or laboratory diagnosis of urinary tract infection (UTI) or reproductive tract infection requiring treatment per current CDC guidelines at screening (may rescreen after treatment).
16. Any condition that, in the opinion of the Principal Investigator or designee, would preclude informed consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving study objectives

Female specific exclusion criteria:

1. Currently pregnant as confirmed by urine HCG test at Screening and Enrollment
2. Currently breastfeeding
3. Intends to become pregnant during the period of study participation
4. Pregnancy outcome 90 days or less prior to Screening
5. Current or planned use of an intravaginal ring
6. Gynecologic or urogenital procedure (e.g., cystoscopy, tubal ligation, dilation and curettage) within 45 days prior to Enrollment (exceptions: IUD insertion/removal, vaginal ultrasound, EMB, biopsy, Pap, colposcopy).
7. Clinically apparent Grade 2 or higher pelvic exam finding (observed by study staff) at Screening or Enrollment.

Note: Cervical bleeding associated with speculum insertion and/or specimen collection judged to be within the range of normal according to the clinical judgment of the IoR/designee is considered expected non-menstrual bleeding and is not exclusionary.

Note: Otherwise, eligible participants with exclusionary pelvic exam findings may be enrolled/randomized after the findings have improved to a non-exclusionary severity grading or resolved within 60 days of providing informed consent for screening.

Male specific exclusion criteria:

1. Diagnosis of phimosis, hypospadias, epispadias, or other abnormality that may impact safety or study evaluations
2. History of treatment for candidal balanoposthitis/balanitis, epididymitis, or other genital lesion (warts, molluscum, etc.) within 30 days prior to Screening
3. Urogenital procedure (e.g., cystoscopy, circumcision, vasectomy) within 45 days prior to enrollment
4. Abnormal semen analysis (sub-study only).
5. Vasectomy (sub-study only)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only cisgender individuals with no history of gender reassignment impacting hormones or genital anatomy are eligible to participate
Enrollment: 72 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | Incidence of treatment-emergent adverse events, measured from first dose through Day 3 post-dose (Lead-in), 21 days post-dose (Phase 1, Stage 1), 28 days post first dose (Phase 1, stage 2) and 24 hours post dose (coital sub-study).
  Number, type, and severity of adverse events observed from first dose through end of follow-up per study section.
Plasma and vaginal fluid concentrations of investigational contraceptive | Time from first dose to last PK sample collection per study section: lead-in up to Day 3; Phase 1 Stage 1 up to Day 21; Phase 1 Stage 2 up to Day 28; sub-study up to 24 hours post dose; samples collected at multiple predefined timepoints.
  Concentrations of the investigational contraceptive measured in blood plasma and vaginal fluid at predefined timepoints from first dose through last PK sample per study section.

SECONDARY OUTCOMES:
Acceptability Questionnaire | Questionnaires administered at Day 2 post-dose during Phase 1, Stage 1 and on the final day of dosing, Day 7 during Phase 1, Stage 2 and immediately after intercourse on Day 3 of the coital sub-study.
  To assess acceptability of IP use
Adherence to dosing schedule | Adherence based on self-reported use evidenced by participant diaries, device logs, or returned product counts post dosing on Day 1 and through Day 7 of the Phase 1, Stage 2 study.
  Adherence to 7-day dosing schedule based on self-reported use evidenced by participant diaries, device logs, or returned product counts

OTHER OUTCOMES:
Anti-viral Activity | Pre and post-dose on Day 1, Day 2 and Day 7 of Phase 1, Stage 1 and after each coital visit during the sub-study.
  To define the relationship between the PK profile of IP and predicted HIV anti-viral activity assessed by TZM-bl assay
Anti-bacterial activity | Pre and post-dose on Day 1, Day 2 and Day 7 of Phase 1, Stage 1 and after each coital visit during the sub-study.
  To define the relationship between the PK profile of IP and predicted Ng anti- bacterial activity assessed by microtitre plate assay
Hyaluronan Binding Assay (HBA) - Vaginal Fluid Exposed to Study Gel (Ex-Vivo) | Pre and post dose day 1, Day 2 and Day 7 of Phase 1, Stage 1
  Proportion of motile, morphologically normal sperm that bind to hyaluronan when applied to vaginal fluid samples that have been collected and then incubated with the study gel ex-vivo (laboratory simulation of product exposure). Samples will be prepared according to validated lab procedures and assessed by light microscopy.
Nugent Score | Pre dose on Day 1 and on Day 7 of Phase 1, Stage 1 and Day 1 and Day 7 of Phase 1, Stage 2
  To assess the impact of IP on vaginal microbiota morphology
Premature acrosomal loss (PAL) assay | After intercourse on Day 2 and Day 3 of the coital sub-study.
  The Premature Acrosomal Loss (PAL) assay evaluates whether exposure to the study product induces premature acrosome exocytosis in human sperm. Sperm samples are incubated with the test article and then stained with a fluorescent acrosome marker (e.g., FITC-PSA or FITC-PNA) to assess acrosomal integrity. The proportion of sperm exhibiting acrosomal loss is quantified by microscopy or flow cytometry and compared with control conditions.
Vaginal Microbiome | Pre-dose on Day 1 and on Day 7 of the Phase 1, Stage 1 and on Day 1, Day 7, Day 14 and Day 21 of Phase 1, stage 2.
  Assessment of the vaginal microbiota using validated culture methods and quantitative PCR (qPCR) assays to detect and quantify key vaginal microbial groups associated with vaginal health.
Vaginal Inflammatory Biomarkers | Pre-dose on Day 1 and Day 7 of Phase 1, Stage 1 and Day 1, Day 7, Day 14 and Day 21 of Phase 1, stage 2.
  Concentrations of selected soluble immune mediators in vaginal fluid, assessed using validated laboratory immunoassays.
Sperm Microscopy (Motility, Morphology, Vitality) | After intercourse on Day 2 and Day 3 of the coital sub-study.
  Sperm microscopy will be performed to assess key semen parameters, including motility, morphology, concentration, and vitality, following WHO laboratory standards.
Eosin-Nigrosin Vitality Stain | After intercourse on Day 2 and Day 3 of the coital sub-study.
  Eosin-Nigrosin (EN) staining will be used to assess sperm viability.
Hyaluronan Binding Assay (HBA) | After intercourse on Day 2 and Day 3 of the coital sub-study.
  The Hyaluronan Binding Assay (HBA) measures the proportion of mature, functionally competent sperm capable of binding to hyaluronan, a component of the cumulus oophorus. Sperm are applied to a hyaluronan-coated slide, and the proportion of motile, morphology-normal sperm that bind is quantified.

CONTACTS AND LOCATIONS:
Overall Officials: Beatrice Chen, MD MPH, Principal Investigator — UPMC Magee-Womens Hospital
Locations (1):
- UPMC Magee-Womens Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
External laboratories will perform assays as part of the study; no plans to share individual participant data outside the study team at this time.